CLINICAL TRIAL: NCT00636168
Title: Adjuvant Immunotherapy With Anti-CTLA-4 Monoclonal Antibody (Ipilimumab) Versus Placebo After Complete Resection of High Risk Stage III Melanoma: A Randomized, Double-blind Phase 3 Trial of the EORTC Melanoma Group
Brief Title: Efficacy Study of Ipilimumab Versus Placebo to Prevent Recurrence After Complete Resection of High Risk Stage III Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA184-029; EORTC 18071
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: High Risk Stage III Melanoma
MeSH Terms: interventions — Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: ipilimumab
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ipilimumab — IV solution, IV, 10 mg/kg, 4x every 21 days, then starting from Week 24 every 12 weeks until Week 156 (3 years), disease recurrence, unacceptable toxicity or patient withdrawal
  Other Names: BMS-734016; MDX-010
  Arms: A
Drug: Placebo — IV solution, IV, 10 mg/kg, 4x every 21 days then starting from Week 24 every 12 weeks until Week 156 (3 years), disease recurrence, unacceptable toxicity or patient withdrawal
  Arms: B

SUMMARY:
The purpose of the study is to determine if ipilimumab is effective in preventing or delaying recurrence and prolongs survival after complete resection of high risk stage III melanoma

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Age ≥ 18 years
* Complete and adequate resection of Stage III melanoma with histologically confirmed melanoma metastatic to lymph node
* Disease-free
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Randomization within 12 weeks of surgery

Exclusion Criteria:

* Prior therapy for melanoma except surgery
* Auto-immune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1211 (Actual)
Dates: Start 2008-06-30 (Actual); Primary Completion 2013-07-26 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (92):
- United States (20):
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - North. Cal. Melanoma Center-St. Mary's Medical Center, San Francisco, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Boca Raton Comprehensive Cancer Center, Boca Raton, Florida
  - H Lee Moffitt Cancer Cnt And Res Inst, Tampa, Florida
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School Of Medicine, St Louis, Missouri
  - Nevada Cancer Center, Las Vegas, Nevada
  - Atlantic Melanoma Center, Morristown, New Jersey
  - University Of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - St Lukes Hospital And Health Network, Bethlehem, Pennsylvania
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee
  - Center For Oncology Research & Treatment, P.A., Dallas, Texas
  - Huntsman Cancer Institute At The Univ. Of Utah, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (7):
  - Local Institution, Waratah, New South Wales
  - Local Institution, Westmead, New South Wales
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Box Hill, Victoria
  - Local Institution, Malvern, Victoria
  - Local Institution, Nedlands, Western Australia
- Austria (2):
  - Local Institution, Graz
  - Local Institution, Vienna
- Belgium (2):
  - Local Institution, Ghent
  - Local Institution, Leuven
- Canada (3):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Montreal, Quebec
- Local Institution, Prague, Czechia
- Denmark (3):
  - Local Institution, Aarhus C
  - Local Institution, Herlev
  - Local Institution, Odense C
- Finland (2):
  - Local Institution, Helsinki
  - Local Institution, Turku
- France (7):
  - Local Institution, Lillie, Cedex
  - Local Institution, Boulogne-Billancourt
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Pierre-Bénite
  - Local Institution, Vandœuvre-lès-Nancy
  - Local Institution, Villejuif
- Germany (10):
  - Local Institution, Berlin
  - Local Institution, Cologne
  - Local Institution, Essen
  - Local Institution, Göttingen
  - Local Institution, Heidelberg
  - Local Institution, Kiel
  - Local Institution, Lübeck
  - Local Institution, Mannheim
  - Local Institution, Tübingen
  - Local Institution, Würzburg
- Italy (6):
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Roma
  - Local Institution, Siena
- Netherlands (4):
  - Local Institution, Amsterdam
  - Local Institution, Leiden
  - Local Institution, Nijmegen
  - Local Institution, Rotterdam
- Local Institution, Oslo, Norway
- Poland (2):
  - Local Institution, Poznan
  - Local Institution, Warsaw
- Russia (12):
  - Local Institution, Pyatigorsk, Stavropol Kray
  - Local Institution, Ivanovo
  - Local Institution, Izhevsk
  - Local Institution, Krasnodar
  - Local Institution, Krasnoyarsk
  - Local Institution, Lipetsk
  - Local Institution, Moscow
  - Local Institution, Petrozavodsk
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Tomsk
  - Local Institution, Ufa
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Zaragoza
- Local Institution, Stockholm, Sweden
- Local Institution, Zurich, Switzerland
- United Kingdom (5):
  - Local Institution, Chelmsford, Essex
  - Local Institution, London, Greater London
  - Local Institution, Southampton, Hampshire
  - Local Institution, Nottingham, Nottinghamshire
  - Local Institution, Leeds, Yorkshire

REFERENCES:
- [Derived] Weber JS, Middleton MR, Yates G, Sharpe DJ, Kurt M, Lobo M, Moshyk A, Vanderpuye-Orgle J, Mohr P. Estimating Long-Term Survivorship Rates Among Patients With Resected Stage III/IV Melanoma: Analyses From CheckMate 238 and European Organization for Research and Treatment of Cancer 18071 Trials. J Clin Oncol. 2025 Mar 10;43(8):929-937. doi: 10.1200/JCO.24.00237. Epub 2024 Oct 8. PMID 39378385
- [Derived] Weber JS, Ascierto PA, Middleton MR, Hennicken D, Zoffoli R, Pieters A, Amadi A, Kupas K, Kotapati S, Moshyk A, Schadendorf D. Indirect treatment comparison of nivolumab versus placebo as adjuvant treatment for resected melanoma. Eur J Cancer. 2021 Nov;158:225-233. doi: 10.1016/j.ejca.2021.08.028. Epub 2021 Oct 15. PMID 34663559
- [Derived] Coens C, Suciu S, Chiarion-Sileni V, Grob JJ, Dummer R, Wolchok JD, Schmidt H, Hamid O, Robert C, Ascierto PA, Richards JM, Lebbe C, Ferraresi V, Smylie M, Weber JS, Maio M, Bottomley A, Kotapati S, de Pril V, Testori A, Eggermont AMM. Health-related quality of life with adjuvant ipilimumab versus placebo after complete resection of high-risk stage III melanoma (EORTC 18071): secondary outcomes of a multinational, randomised, double-blind, phase 3 trial. Lancet Oncol. 2017 Mar;18(3):393-403. doi: 10.1016/S1470-2045(17)30015-3. Epub 2017 Feb 3. PMID 28162999
- [Derived] Eggermont AM, Chiarion-Sileni V, Grob JJ, Dummer R, Wolchok JD, Schmidt H, Hamid O, Robert C, Ascierto PA, Richards JM, Lebbe C, Ferraresi V, Smylie M, Weber JS, Maio M, Bastholt L, Mortier L, Thomas L, Tahir S, Hauschild A, Hassel JC, Hodi FS, Taitt C, de Pril V, de Schaetzen G, Suciu S, Testori A. Prolonged Survival in Stage III Melanoma with Ipilimumab Adjuvant Therapy. N Engl J Med. 2016 Nov 10;375(19):1845-1855. doi: 10.1056/NEJMoa1611299. Epub 2016 Oct 7. PMID 27717298
- [Derived] Eggermont AM, Chiarion-Sileni V, Grob JJ, Dummer R, Wolchok JD, Schmidt H, Hamid O, Robert C, Ascierto PA, Richards JM, Lebbe C, Ferraresi V, Smylie M, Weber JS, Maio M, Konto C, Hoos A, de Pril V, Gurunath RK, de Schaetzen G, Suciu S, Testori A. Adjuvant ipilimumab versus placebo after complete resection of high-risk stage III melanoma (EORTC 18071): a randomised, double-blind, phase 3 trial. Lancet Oncol. 2015 May;16(5):522-30. doi: 10.1016/S1470-2045(15)70122-1. Epub 2015 Mar 31. PMID 25840693
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol definition of Enrolled population: All 1211 participants who signed the Informed Consent Form; 951 were randomized to treatment and 945 were treated. Reasons for not being randomized: 193 were ineligible; 42 refused; 19 could not be randomized within 12 weeks after complete lymph node dissection; 6 due to other reasons.
Groups:
- Ipilimumab 10mg/kg: Ipilimumab (10 mg/kg) as a single dose via a 90 minute intravenous (IV) infusion (not as bolus or IV push) during Days 1, 22, 43 and 64 (every 21 days in the Induction Phase) for a total of four separate doses, until disease recurrence, unacceptable toxicity or withdrawal of consent. During the maintenance phase, Ipilimumab was administered at a dose of 10 mg/kg, by IV infusion, every 12 weeks, beginning at Week 24, until disease recurrence, unacceptable toxicity or withdrawal of consent, for a maximum of 3 years (Week 156).
- Placebo: Placebo as a single dose via a 90 minute intravenous (IV) infusion (not as bolus or IV push) during Days 1, 22, 43 and 64 (Induction Phase) for a total of four separate doses, until disease recurrence, unacceptable toxicity or withdrawal of consent. During the maintenance phase, placebo was administered by IV infusion every 12 weeks, beginning at Week 24, until disease recurrence, unacceptable toxicity or withdrawal of consent, for a maximum of 3 years (Week 156).
Period: Randomized to Study Drug
Arm/Group | Ipilimumab 10mg/kg | Placebo
Started | 475 | 476
Completed | 471 | 474
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — No longer meets study criteria | 1 | 0
Period: Treated With Study Drug
Arm/Group | Ipilimumab 10mg/kg | Placebo
Started | 471 | 474
Completed (Normal Completion) | 63 | 143
Not Completed | 408 | 331
Not completed — Recurrence of disease | 135 | 282
Not completed — Adverse Event | 250 | 22
Not completed — Participant withdrew consent | 16 | 21
Not completed — Poor/non-compliance | 1 | 3
Not completed — Death | 3 | 0
Not completed — Pregnancy | 1 | 0
Not completed — No longer meets study criteria | 1 | 0
Not completed — Other reason | 1 | 3
Period: Long Term Follow-Up
Arm/Group | Ipilimumab 10mg/kg | Placebo
Started (Continuing in Long Term Follow Up) | 141 | 143
Completed | 130 | 129
Not Completed | 11 | 14
Not completed — Lost to Follow-up | 3 | 3
Not completed — Participant withdrew consent | 0 | 2
Not completed — Death | 8 | 9

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants, analyzed in the arm to which they were allocated by randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab 10mg/kg | Placebo | Total
Number analyzed (Participants) | 475 | 476 | 951
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (12.90) | 51.5 (12.82) | 51.1 (12.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 183 | 362
  Male | 296 | 293 | 589
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 470 | 476 | 946
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Free Survival (RFS) Per Independent Review Committee (IRC) in the Intent to Treat (ITT) Population
Description: Recurrence free survival (RFS) was programmatically determined based on the disease recurrence data provided by the IRC and was defined as the time between the date of randomization and the date of first recurrence or death (whatever the cause), whichever occurred first. A participant who died without reported recurrence was considered to have recurrence on the date of death. For those participants who remained alive and recurrence-free, RFS was censored on the date of last evaluable post-randomization tumor assessment. For those who remained alive and had no recorded post-randomization tumor assessment, RFS was censored on the day of randomization. Participants with disease at baseline were considered to have an event on the day of randomization. Computerized tomography (CT) and magnetic resonance imaging (MRI) were mandatory to establish recurrence. The primary analysis was event-driven and planned when at least 512 RFS events assessed per IRC were collected.
Time Frame: Date of randomization to first date of recurrence or death or last available disease assessment with RFS data up to 5 years. Median follow-up was 2.7 years.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab 10mg/kg | Placebo
Number analyzed (Participants) | 475 | 476
months | 26.09 [19.32 to 39.26] | 17.05 [13.40 to 21.62]
Statistical Analysis 1: Comparison: Ipilimumab 10mg/kg vs Placebo; The hazard ratio, and its 95 % confidence interval was estimated using a Cox proportional hazards model, stratified by stage (IIIa vs. IIIb vs. IIIc with 1-3 positive lymph-nodes vs. IIIc with >= 4 positive lymph-nodes) as indicated at randomization, with treatment as the single covariate.. The analysis was performed after 528 RFS events per IRC were reported. Two-sided, 95% confidence intervals for median RFS were computed by the Brookmeyer and Crowley method using log-log transformation; Test type: Superiority; p = 0.0013, Log Rank; stratified 2-sided log-rank test; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.64 to 0.90]

2. Primary Outcome: Number of Participants With Recurrence or Death as Per Independent Review Committee (IRC) in the Intent to Treat (ITT) Population
Description: Recurrence was defined as appearance of one or more new melanoma lesions: local, regional or distant metastasis. Computerized tomography (CT) and magnetic resonance imaging (MRI) were mandatory to establish recurrence. A participant who died without reported recurrence was considered to have recurred on the date of death. Disease was assessed at randomization and every 12 weeks (±2 weeks) for 3 years, then every 24 weeks until documented distant progression.
Time Frame: Date of randomization to first date of recurrence or death or last available disease assessment with RFS data upto 5 years. Median follow-up was 2.7 years.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab 10mg/kg | Placebo
Number analyzed (Participants) | 475 | 476
Participants | 234 [19.32 to 39.26] | 294 [13.40 to 21.62]

3. Primary Outcome: Recurrence-Free Survival (RFS) Rates Per IRC at 1 Year, 2 Years, and 3 Years in the ITT Population
Description: Yearly recurrence-free survival rates, eg. at 1 year, defined as the probability that a participant was recurrence-free at 1 year following randomization, were estimated for each treatment group using the Kaplan-Meier product-limit method, along with their corresponding log-log transformed 95% confidence intervals. RFS was defined as the time between the date of randomization and the date of first recurrence or death (whatever the cause), whichever occurred first. A participant who died without reported recurrence was considered to have recurrence on the date of death. For those who remained alive and recurrence-free, RFS was censored on the date of last evaluable post-randomization tumor assessment. For those who remained alive and had no recorded post-randomization tumor assessment, RFS was censored on the day of randomization. Participants with disease at baseline were considered to have an event on the day of randomization. CT and MRI were mandatory to establish recurrence.
Time Frame: At years 1, 2, and 3
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab 10mg/kg | Placebo
Number analyzed (Participants) | 475 | 476
Percentage of participants
  RFS Rate at 1 Year | 63.50 [58.89 to 67.74] | 56.13 [51.52 to 60.47]
  RFS Rate at 2 Years | 51.45 [46.69 to 56.00] | 43.83 [39.27 to 48.28]
  RFS Rate at 3 Years | 46.48 [41.46 to 51.34] | 34.79 [30.12 to 39.50]

4. Secondary Outcome: Distant Metastasis-Free Survival (DMFS) Per Independent Review Committee (IRC) in the Intent to Treat (ITT) Population
Description: Distant Metastasis-Free Survival (DMFS) was programmatically determined based on the first date of distant metastasis provided by the IRC and was defined as the time between the date of randomization and the date of first distant metastasis or death (whatever the cause), whichever occurred first. A participant who died without reported disease distant metastasis was considered to have distant metastasis on the date of death. For those who remained alive and metastasis-free, DMFS was censored on the date of last evaluable post-randomization tumor assessment. For those who remained alive and had no recorded post-randomization tumor assessment, DMFS was censored on the day of randomization. Participants with disease at baseline were considered to have an event on the day of randomization. Disease was assessed at baseline (randomization) and every 12 weeks (±2 weeks) for 3 years, then every 24 weeks until documented distant progression.
Time Frame: From June 2008 to January 2016 (approximately 90 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab 10mg/kg | Placebo
Number analyzed (Participants) | 475 | 476
Months | 48.30 [35.45 to 71.56] | 27.47 [21.91 to 34.79]
Statistical Analysis 1: Comparison: Ipilimumab 10mg/kg vs Placebo; Medians and associated 2-sided 95% confidence intervals are calculated using the method of Brookmeyer and Crowley. Analysis was stratified for stage (IIIa vs. IIIb vs. IIIc with 1-3 positive lymph-nodes vs. IIIc with >= 4 positive lymph-nodes) as recorded at randomization. P-value was based on stratified 2-sided log-rank test. Hazard of 10 mg/kg Ipilimumab over hazard of Placebo, with 2-sided 95.8% confidence interval are based on a stratified Cox proportional hazards model; Test type: Superiority; p = 0.0024, Log Rank; stratified 2-sided log-rank test; Hazard Ratio (HR) = 0.76, 95.8% CI 2-sided [0.64 to 0.92]

5. Secondary Outcome: Number of Participants With Distant Metastasis-Free Survival (DMFS) Per Independent Review Committee (IRC) in the Intent to Treat (ITT) Population
Description: DMFS was programmatically determined based on the first date of distant metastasis provided by the IRC and was defined as the time between the date of randomization and the date of first distant metastasis or death (whatever the cause), whichever occurred first. A participant who died without reported disease distant metastasis was considered to have distant metastasis on the date of death. For those who remained alive and metastasis-free, DMFS was censored on the date of last evaluable post-randomization tumor assessment. For those who remained alive and had no recorded post-randomization tumor assessment, DMFS was censored on the day of randomization. Participants with disease at baseline were considered to have an event on the day of randomization. Disease was assessed at baseline (randomization) and every 12 weeks (2 weeks) for 3 years, then every 24 weeks until documented distant progression.
Time Frame: From June 2008 to January 2016 (approximately 90 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab 10mg/kg | Placebo
Number analyzed (Participants) | 475 | 476
Participants | 227 | 279

6. Secondary Outcome: Distant Metastasis-Free Survival (DMFS) Rates Per IRC at 1 Year, 2 Years, 3 Years, 4 Years and 5 Years in the ITT Population
Description: Yearly distant metastasis-free survival rates, e.g. at 1 year, defined as the probability that a participant was alive at 1 year following randomization, were estimated via the Kaplan-Meier method. Distant Metastasis-Free Survival (DMFS) was programmatically determined based on the first date of distant metastasis provided by the IRC and was defined as the time between the date of randomization and the date of first distant metastasis or death (whatever the cause), whichever occurred first. A participant who died without reported disease distant metastasis was considered to have distant metastasis on the date of death. For those who remained alive and metastasis-free, DMFS was censored on the date of last evaluable post-randomization tumor assessment. For those who remained alive and had no recorded post-randomization tumor assessment. Participants with disease at baseline were considered to have an event on the day of randomization.
Time Frame: At years 1, 2, 3, 4 and 5
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab 10mg/kg | Placebo
Number analyzed (Participants) | 475 | 476
Percentage of participants
  DMFS Rate at 1 Year | 74.27 [69.98 to 78.04] | 65.77 [61.27 to 69.88]
  DMFS Rate at 2 Years | 61.48 [56.75 to 65.85] | 53.26 [48.58 to 57.70]
  DMFS Rate at 3 Years | 53.90 [49.04 to 58.50] | 45.17 [40.53 to 49.70]
  DMFS Rate at 4 Years | 50.19 [45.30 to 54.87] | 41.48 [36.87 to 46.02]
  DMFS Rate at 5 Years | 48.29 [43.36 to 53.04] | 38.90 [34.29 to 43.47]

7. Secondary Outcome: Overall Survival in the Intent to Treat (ITT) Population
Description: OS was defined as the time from the date of randomization to the date of death. For those participants who had not died, OS was censored at the recorded last non-missing date of contact for which the participant was known to be alive.
Time Frame: From June 2008 to January 2016 (approximately 90 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab 10mg/kg | Placebo
Number analyzed (Participants) | 475 | 476
Months | 86.60 [86.60 to NA] — Upper limit was not reached because the number of participants with a followup of more than 7 years was too small | NA [59.30 to NA] — Median and upper limit were not reached because the number of participants with a followup of more than 7 years was too small
Statistical Analysis 1: Comparison: Ipilimumab 10mg/kg vs Placebo; Medians and associated 2-sided 95% confidence intervals are calculated using the method of Brookmeyer and Crowley. Analysis was stratified for stage (IIIa vs. IIIb vs. IIIc with 1-3 positive lymph-nodes vs. IIIc with >= 4 positive lymph-nodes) as recorded at randomization. P-value was based on stratified 2-sided log-rank test. Hazard of 10 mg/kg Ipilimumab over hazard of Placebo, with 2-sided 95.1% confidence interval are based on a stratified Cox proportional hazards model; Test type: Superiority; p = 0.0013, Log Rank; stratified 2-sided log-rank test; Hazard Ratio (HR) = 0.72, 95.1% CI 2-sided [0.58 to 0.88]

8. Secondary Outcome: Rate of Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death. For those participants who had not died, OS was censored at the recorded last non-missing date of contact for which the participant was known to be alive.Yearly survival rates, e.g. at 3 years, defined as the probability that a participant was alive at 3 years following randomization, were estimated via the Kaplan-Meier method
Time Frame: From date of randomization to date of death, assessed up to 9 years
Population: Intent to Treat Population: All randomized participants,analyzed in the arm to which they were allocated by randomization
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab 10mg/kg | Placebo
Number analyzed (Participants) | 475 | 476
Percentage of participants
  OS Rate at 1 year | 93.53 [90.88 to 95.43] | 87.72 [84.40 to 90.37]
  OS Rate at 2 years | 82.55 [78.76 to 85.73] | 75.27 [71.10 to 78.92]
  OS Rate at 3 years | 74.20 [69.90 to 77.98] | 65.43 [60.91 to 69.56]
  OS Rate at 4 years | 67.79 [63.24 to 71.90] | 60.34 [55.72 to 64.64]
  OS Rate at 5 years | 65.42 [60.80 to 69.64] | 54.43 [49.71 to 58.89]
  OS Rate at 7 years | 60.0 [55.0 to 64.7] | 51.3 [46.5 to 55.9]

9. Secondary Outcome: Number of Participants With On-Study Adverse Events (AEs) Leading to Discontinuation of Treatment, Serious AEs (SAEs), Drug-Related SAEs, Immune-related AEs (irAEs), Immune-mediated Adverse Reactions (imARs), Deaths in Treated Population
Description: AEs: Medical Dictionary for Regulatory Activities (MedDRA) version 16.1. irAEs=unknown etiology consistent with an immune phenomenon, considered as causally related to drug. imARs=based on investigator's assessment of immune-mediated etiology [excluding novel maintenance events (ie, patients with imARs occurring for the first time during maintenance)]. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Drug-related (D-R)=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling, Gr 5=Death.
Time Frame: Day 1 up to 70 days after last dose; up to 5 years
Population: Safety population: All randomized participants who received at least 1 dose of study therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab 10mg/kg | Placebo
Number analyzed (Participants) | 471 | 474
Participants
  On-study AE leading to Discontinuation (Any Grade) | 247 | 43
  On-study SAE (At least 5%, Any Grade) | 257 | 128
  On-study D-R SAE (Any Grade) | 217 | 10
  On-study irAE (Any Grade) | 426 | 188
  On-study gastrointestinal irAE (Any Grade) | 217 | 85
  On-study endocrine irAE (Any Grade) | 178 | 38
  On-study liver irAE (Any Grade) | 115 | 20
  On-study skin irAE (Any Grade) | 298 | 99
  On-study neurological irAE (Any Grade) | 21 | 9
  On-study other irAE (Any Grade) | 111 | 23
  On-study imAR (Grade 3-4) | 194 | 16
  On-study imAR (Grade 5) | 1 | 0
  On-study enterocolitis imAR (Grade 5) | 1 | 0
  On-study enterocolitis imAR (Grade 3-4) | 76 | 4
  On-study endocrinopathy imAR (Grade 3-4) | 39 | 1
  On-study hepatitis imAR (Grade 3-4) | 51 | 1
  On-study dermatitis imAR (Grade 3-4) | 19 | 2
  On-study neuropathy imAR (Grade 3-4) | 10 | 0
  On-study other imAR (Grade 3-4) | 30 | 9
  Any Death | 162 | 214
  Death within 70 days of last dose study drug | 6 | 6
  Death within 30 days of last dose study drug | 1 | 0
  Drug-related Deaths | 4 | 0

10. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Non-serious AEs (NSAEs) and Number of Deaths: Overall Study
Description: AEs: Medical Dictionary for Regulatory Activities (MedDRA) version 16.1. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: SAEs and NSAEs: Day 1 up to 70 days after last dose(safety window). Deaths: All deaths regardless of 70 day safety window.Up to 10 years
Population: Safety population: All randomized participants who received at least 1 dose of study therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab 10mg/kg | Placebo
Number analyzed (Participants) | 471 | 474
Participants
  No. of deaths | 173 | 223
  No. of participants with SAEs | 257 | 128
  No of participants with NSAEs | 441 | 382

11. Secondary Outcome: Exposure Adjusted Incidence Rate of Adverse Events Including Multiple Occurrences of Unique Events
Description: P-Y = person-years of exposure. Incidence rate per 100 person-years of exposure (IR/100 P-Y) was calculated as event count * 100 /person-years of exposure. MedDRA Version: 19. Duplicate AEs have been eliminated and overlapping and contiguous occurrences of the same event have been collapsed.
Time Frame: Day 1 up to 70 days after last dose; up to 5 years
Population: All participants who received at least one dose of ipilimumab or placebo, adjusted for person-years (P-Y) of exposure; P-Y=467.4; P-Y=781.7 for ipilimumab and placebo, respectively.
Measure: Number; unit: Events per 100 person-years of exposure
Arm/Group | Ipilimumab 10mg/kg | Placebo
Number analyzed (Participants) | 471 | 474
Events per 100 person-years of exposure | 1171.8 | 465.0

12. Secondary Outcome: Mean Change From Baseline in Global Health Status Scores at Each Assessment Timepoint
Description: Global health status was measured using European Organization for Research and Treatment of Cancer (EORTC) Quality Life Questionnaire (QLQ) C-30. This health related quality of life (HRQoL) questionnaire was comprised of 15 questions on functional scales, 13 questions on symptom scales and 2 on global health status scale. Global Health Status used a 7 point Likert-type scale of 1 (Very poor) to 7 (Excellent). All scales linearly transformed to 0-100 scales. Higher scores for Global Health Status indicate better HRQoL. An increase from baseline indicates improvement in HRQoL compared to baseline. HRQoL was administered within 1 week prior to first dose (baseline) and on Days 22, 43, 64 (+/- 3 days), Week 24 and every 12 weeks up to 2 years, independent of disease progression.
Time Frame: Baseline up to 2 years from randomization
Population: All randomized participants (ITT) analyzed in the arm to which they were allocated by randomization were analyzed. At timepoint level, all randomized participants (ITT) with a measurement at the timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ipilimumab 10mg/kg | Placebo
Number analyzed (Participants) | 400 | 421
units on a scale
  Week 4 Day 22 | -2.29 (15.96) | 1.33 (14.02)
  Week 7, Day 43: number analyzed (Participants) | 360 | 412
  Week 7, Day 43 | -6.64 (20.44) | -0.10 (16.75)
  Week 10 Day 64: number analyzed (Participants) | 356 | 405
  Week 10 Day 64 | -9.06 (23.56) | -0.23 (16.18)
  Week 24 Day 162 (300, 347): number analyzed (Participants) | 300 | 347
  Week 24 Day 162 (300, 347) | -4.33 (21.55) | 1.37 (17.00)
  Week 36 Day 246: number analyzed (Participants) | 290 | 307
  Week 36 Day 246 | -5.09 (21.32) | 1.52 (18.52)
  Week 48 Day 330: number analyzed (Participants) | 275 | 276
  Week 48 Day 330 | -3.67 (20.17) | 1.54 (18.87)
  Week 60 Day 414: number analyzed (Participants) | 242 | 255
  Week 60 Day 414 | -5.30 (21.34) | 2.84 (17.05)
  Week 72 day 498: number analyzed (Participants) | 217 | 248
  Week 72 day 498 | -4.07 (23.19) | 1.18 (17.46)
  Week 84 Day 582: number analyzed (Participants) | 205 | 227
  Week 84 Day 582 | -3.90 (22.06) | 1.84 (17.08)
  Week 96 Day 666: number analyzed (Participants) | 199 | 214
  Week 96 Day 666 | -4.48 (21.71) | 1.36 (18.67)
  Week 108 Day 750: number analyzed (Participants) | 162 | 177
  Week 108 Day 750 | -4.27 (20.35) | 2.45 (16.72)

ADVERSE EVENTS:
Time Frame: Day 1 up to 70 days after last dose. Up to 10 years.
Description: Adverse Events were collected for the safety population which included all 945 randomized subjects who received at least 1 dose of study therapy (471 in the ipilimumab group and 474 in the placebo group)
Arm/Group | IPILIMUMAB 10 MG/KG | PLACEBO
All-Cause Mortality (participants affected / at risk) | 173/471 | 223/474
Serious Adverse Events (participants affected / at risk) | 257/471 | 128/474
Other Adverse Events (participants affected / at risk) | 441/471 | 382/474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IPILIMUMAB 10 MG/KG (N=471) | PLACEBO (N=474)
Lymphadenopathy (Blood and lymphatic system disorders) | 5 | 3
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Bifascicular block (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Silent myocardial infarction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 4 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Basedow's disease (Endocrine disorders) | 1 | 0
Endocrine disorder (Endocrine disorders) | 1 | 1
Hyperadrenocorticism (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 37 | 0
Hypopituitarism (Endocrine disorders) | 10 | 0
Hypothyroidism (Endocrine disorders) | 3 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 5 | 0
Thyroiditis (Endocrine disorders) | 1 | 0
Autoimmune uveitis (Eye disorders) | 1 | 0
Episcleritis (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 4 | 0
Colitis (Gastrointestinal disorders) | 51 | 1
Colitis ulcerative (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 36 | 6
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 2
Intestinal perforation (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 1
Adverse event (General disorders) | 1 | 0
Asthenia (General disorders) | 3 | 0
Chest pain (General disorders) | 3 | 2
Disease progression (General disorders) | 1 | 4
Disease recurrence (General disorders) | 0 | 3
Fatigue (General disorders) | 5 | 1
Influenza like illness (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pyrexia (General disorders) | 18 | 1
Retention cyst (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 12 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 4 | 0
Hepatocellular injury (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 5 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Anaphylactoid reaction (Immune system disorders) | 1 | 0
Autoimmune disorder (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 3 | 0
Sarcoidosis (Immune system disorders) | 3 | 1
Appendicitis (Infections and infestations) | 3 | 1
Appendicitis perforated (Infections and infestations) | 0 | 3
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 4
Cystitis (Infections and infestations) | 3 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 2 | 7
External ear cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Groin infection (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0
Herpes ophthalmic (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 2 | 0
Meningitis aseptic (Infections and infestations) | 2 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1
Neuroborreliosis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Septic embolus (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 2 | 0
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Respiratory tract procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 17 | 0
Aspartate aminotransferase increased (Investigations) | 15 | 0
Blood corticotrophin decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Influenza A virus test positive (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Lymph nodes scan abnormal (Investigations) | 1 | 1
Thyroid function test abnormal (Investigations) | 2 | 0
Transaminases increased (Investigations) | 3 | 0
Weight decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 12
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endobronchial lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 9
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 7
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 11
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Ataxia (Nervous system disorders) | 0 | 1
Autoimmune neuropathy (Nervous system disorders) | 1 | 0
Axonal neuropathy (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral thrombosis (Nervous system disorders) | 0 | 1
Cranial nerve disorder (Nervous system disorders) | 1 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 2
Meningoradiculitis (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 2
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Trigeminal nerve disorder (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 4 | 0
Lymphoedema (Vascular disorders) | 1 | 1
Withdrawal hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IPILIMUMAB 10 MG/KG (N=471) | PLACEBO (N=474)
Hypophysitis (Endocrine disorders) | 56 | 2
Hypothyroidism (Endocrine disorders) | 47 | 7
Abdominal pain (Gastrointestinal disorders) | 64 | 44
Colitis (Gastrointestinal disorders) | 43 | 5
Constipation (Gastrointestinal disorders) | 31 | 30
Diarrhoea (Gastrointestinal disorders) | 229 | 141
Nausea (Gastrointestinal disorders) | 117 | 82
Vomiting (Gastrointestinal disorders) | 61 | 27
Asthenia (General disorders) | 29 | 38
Fatigue (General disorders) | 188 | 143
Influenza like illness (General disorders) | 35 | 30
Oedema peripheral (General disorders) | 21 | 27
Pyrexia (General disorders) | 73 | 22
Nasopharyngitis (Infections and infestations) | 21 | 31
Alanine aminotransferase increased (Investigations) | 95 | 26
Aspartate aminotransferase increased (Investigations) | 72 | 26
Blood lactate dehydrogenase increased (Investigations) | 33 | 12
Blood testosterone decreased (Investigations) | 29 | 8
Lipase increased (Investigations) | 42 | 30
Weight decreased (Investigations) | 149 | 42
Weight increased (Investigations) | 71 | 114
Decreased appetite (Metabolism and nutrition disorders) | 65 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 45
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 41
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 | 26
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 36
Dizziness (Nervous system disorders) | 29 | 18
Headache (Nervous system disorders) | 150 | 85
Anxiety (Psychiatric disorders) | 21 | 25
Insomnia (Psychiatric disorders) | 45 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 68 | 48
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 16
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 26 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 203 | 70
Rash (Skin and subcutaneous tissue disorders) | 186 | 80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.